CLINICAL TRIAL: NCT03669315
Title: Modulating Inhibitory Control Networks in Gambling Disorder With Theta Burst Stimulation
Acronym: TMS-GD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CNS Onlus (Other)
Responsible Party: Principal Investigator, Stefano Pallanti, Professor, CNS Onlus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS-GD
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Gambling Disorder
Keywords: Gambling Disorder; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Gambling | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: After selection and enrollment, participants will be screened at baseline with MRI and a complete diagnostic and clinical assessment, described in the following corresponding sections. Using a placebo-controlled double-blind design patients will be randomized to receive active or placebo cTBS.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Outcome assessor, investigators and participants will be blinded to the type of treatment (active TMS or Placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active cTBS treatment (Active Comparator): Active cTBS will be administered with a Magventure MagPro Stimulator R30 using a butterfly coil. TBS consists of bursts of 3 pulses separated by 20ms (i.e. 50 Hz), with each triplet being repeated every 200 ms (i.e. 5 Hz). Stimulus intensities will be set at 80% of AMT. The investigators will use 2 trains of 600 pulses each separated by 1 minute (a total of 1200 pulses).
  Interventions: Device: Transcranial Magnetic stimulation
- Sham cTBS treatment (Sham Comparator): Sham cTBS will be administered with a Magventure MagPro Stimulator R30 using a butterfly sham coil. The same active cTBS configuration will be used.
  Interventions: Device: Transcranial Magnetic stimulation

INTERVENTIONS:
Device: Transcranial Magnetic stimulation — Neuromodulation tool

SUMMARY:
In this project the investigators propose a randomized double-blind placebo-controlled design in which 40 patients with GD will receive active or sham cTBS to the pre-SMA for 2 weeks. The investigators will combine TMS, multimodal structural and functional MRI and behavioral measures in order to identify circuit-level mechanisms of action and therapeutic targets (connectivity changes that explain clinical improvement) and assess the efficacy of TMS in modulating inhibitory control and symptom severity in this population.

DETAILED DESCRIPTION:
SPECIFIC AIMS The appropriate interplay of cognitive and reward systems is essential for adaptive human behavior, allowing a homeostatic balance between immediate basic pleasures and long-term planned rewards. Deficits in inhibitory control from cortical cognitive systems over subcortical reward circuits is a key pathophysiological feature of addictive behavior that has not been studied satisfactorily in gambling disorder (GD). The clinical phenotype of this population is characterized by unsuccessful efforts to reduce or stop gambling despite negative outcomes, suggestive of faulty inhibitory control of gambling impulses that sustain the chronicity and comorbidities of this clinical syndrome. Deficits in behavioral and cognitive control constitute a symptom dimension associated with diminished response inhibition in experimental tasks such as the Stop Signal Task (SST). The pre-supplementary motor area (pre-SMA) is a key node of the cognitive control network responsible for response inhibition. Pre-SMA activation has been associated to response inhibition performance in fMRI studies using the SST and recent evidence also suggests that its activity represents a motivational signal for movement. In fact, pre-SMA seems to have a dominant role in bridging the delay between expected reward and specific actions rather than determining whether an action is made. Although the pathophysiology of GD is not well understood, studies have shown altered brain activity in prefrontal regions (including pre-SMA) of GD patients during response inhibition tasks in addition to functional connectivity abnormalities of SMA during rest. These circuit-level abnormalities represent a potential therapeutic target that could be modulated by brain stimulation therapies such as transcranial magnetic stimulation (TMS). Theta burst stimulation (TBS), is a particularly brief and effective form of TMS that can be inhibitory (continuous or cTBS) or excitatory (intermittent or iTBS). Although pre-SMA has been successfully targeted with traditional TMS and TBS for impulse-control disorders like OCD, this approach has never been tested for GD in therapeutic or mechanistic studies. Despite the significant morbidity and mortality of GD, there is a dramatic shortage of effective treatment options for these patients, partly due to the lack of valid pathophysiological models for target discovery and experimental therapeutics. In this project the investigators propose a randomized double-blind placebo-controlled design in which 40 patients with GD will receive active or sham cTBS to the pre-SMA for 2 weeks. The investigators will combine TMS, multimodal structural and functional MRI and behavioral measures in order to identify circuit-level mechanisms of action and therapeutic targets (connectivity changes that explain clinical improvement) and assess the efficacy of TMS in modulating inhibitory control and symptom severity in this population.

Aim 1 (ACUTE MECHANISM OF ACTION): To assess circuit-level effects of a single session of cTBS to the pre-SMA in GD patients. Hypothesis 1.1: cTBS will lead to increase in functional connectivity between cortical inhibitory nodes (pre-SMA) and reward subcortical structures (Nucleus Accumbens, NAc), and these changes will correlate with improvement in reaction time in SST. Hypothesis 1.2: cTBS will not lead to acute changes in FA, RD or AD in the mesocorticolimbic pathway. Hypothesis 1.3: cTBS will lead to increased cognitive control network and decreased NAc activation during SST. Exploratory analyses will test the predictive value of acute circuit changes for clinical improvement after 2 weeks and 1 month follow up.

Aim 2 (CHRONIC MECHANISM OF ACTION): To assess circuit-level effects of 10 session of cTBS to the pre-SMA in GD patients Hypothesis 2.1: cTBS will lead to increases in functional connectivity between preSMA and NAc, and these will correlate with behavioral and clinical improvement. Hypothesis 2.2: cTBS will lead to increased FA and decreased RD and AD in the mesocorticolimbic pathway, and these will correlate with clinical improvement. Hypothesis 2.3: cTBS will lead to further increased cognitive control network and decreased NAc activation during SST, and these will correlate with clinical improvement.

Aim 3 (BEHAVIORAL/CLINICAL): To determine the behavioral and clinical changes of cTBS to the preSMA in GD. Hypothesis 3.1: A single session of cTBS will lead to improvement in reaction time in the SST, but not in symptom severity measured with clinical scales. Hypothesis 3.2: 10 sessions of cTBS will lead to improvement in reaction time in the behavioral inhibition task, in addition to a reduction in clinical severity (including craving/urges) as measured by clinical scales.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of Gambling Disorder
2. Age between 18 and 65 years

Exclusion Criteria:

1. any additional current psychiatric comorbidity, except for nicotine addiction;
2. a lifetime DSM-5 diagnosis of schizophrenia or other psychotic syndromes, substance dependence or substance abuse, including alcohol, bipolar I or II disorder, mental disorder due to a general medical condition;
3. serious suicide risk;
4. illness duration less than two years;
5. hospitalization in the last 6 months;
6. the inability to receive TMS because of metallic implants, or history of seizures (personal or family history of seizure in first degree relatives);
7. any major medical disease;
8. pregnancy or nursing of an infant;
9. the inability or refusal to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
cTBS effects on gambling symptoms change | Baseline - Day 10 (after 10 cTBS sessions) - after 1 month follow-up
  cTBS effects on gabling symptoms severity assessed through the PG-Y-BOCS (Yale-Brown Obsessive-Compulsive Scale modified for Pathological Gambling). Range from: 0-40 (higher values=worse symptoms)
cTBS effects on gambling symptoms change | Baseline - Day 10 (after 10 cTBS sessions) - after 1 month follow-up
  cTBS effects on gabling symptoms severity assessed through the GUQ (Gambling Urges Questionnaire). Range from: 0-60 (higher values=worse symptoms)

SECONDARY OUTCOMES:
Acute mechanism of action | Day 1
  Functional MRI assessment
Chronic mechanism of action | Day 10
  Functional MRI assessment

CONTACTS AND LOCATIONS:
Locations (1):
- CNSOnlus, Institute of Neuroscience, Florence, Italy

IPD SHARING:
Plan to Share IPD: No